CLINICAL TRIAL: NCT06977074
Title: Prospective Phase II Proof-of-Concept Trial on Circulating Tumor DNA (ctDNA)-Optimized Induction Immunochemotherapy Cycle Reduction for Resectable Non-Small Cell Lung Cancer
Brief Title: PROPHET Study: ctDNA-Guided Personalized Induction Immunochemotherapy for NSCLC
Acronym: PROPHET
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Ze-Rui Zhao, Dr. Ze-Rui Zhao, Sun Yat-sen University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: B2025-176-01
Record Dates: First submitted 2025-05-01; First posted 2025-05-16 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Non-small Cell Lung Cancer (NSCLC)
Keywords: Non-small cell lung cancer; ctDNA; Induction therapy; Immunochemotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Immune Checkpoint Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Induction immunochemotherapy (Experimental)
  Interventions: Drug: PD-1 inhibitor; Drug: Platinum Doublet

INTERVENTIONS:
Drug: PD-1 inhibitor — Two to four cycles of tislelizumab at a dose of 200 mg every three weeks, along with a platinum-based chemotherapy doublet based on the result of ctDNA dynamics
Drug: Platinum Doublet — Platinum-based chemotherapy (carboplatin AUC=5 + pemetrexed 500 mg/m² [adenocarcinoma] or nab-paclitaxel 260 mg/m² [squamous/other subtypes])

SUMMARY:
The goal of this clinical trial is to evaluate the clinical value of ctDNA testing in guiding the optimization of immunochemotherapy cycles during induction treatment for resectable patients with NSCLC. The main questions it aims to answer are:

* Does ctDNA clearance indicate pathological complete response?
* Are additional cycles of immunochemotherapy necessary for patients who have ctDNA clearance after initial cycles of treatment? Researchers will use ctDNA dynamics to guide the cycles of induction treatment to see if some patients can avoid excessive cycles of treatment.

DETAILED DESCRIPTION:
Advances in precision medicine have highlighted the potential of circulating tumor DNA (ctDNA) detection in NSCLC diagnosis, treatment efficacy monitoring, and prognosis evaluation. Induction immunotherapy combined with chemotherapy is now a standard treatment for patients with resectable NSCLC, but optimizing the number of immunochemotherapy cycles to enhance efficacy and reduce toxicity remains a critical clinical challenge. In this Phase II, proof-of-concept trial, around 83 patients with AJCC stage IIA-IIIB NSCLCs who are deemed resectable by an MDT team will participate to evaluate the potential role of dynamic ctDNA changes in guiding the cycle reduction of induction immunotherapy combined with chemotherapy while maintaining overall efficacy.

Eligible patients will receive 2 cycles (21-day intervals) of PD-1 inhibitor + platinum-based chemotherapy. Subsequent cycles (1-2 additional cycles) are determined by ctDNA status via tumour-agnostic strategies:

1. For patients with ctDNA clearance: Randomized (1:1) to surgery or continued therapy.
2. For patients with ctDNA persistence: Sequential 1-2 additional cycles. For all patients who are available to undergo surgery, the operation will be performed 4-6 weeks following the last cycle of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically/cytologically confirmed, untreated stage IIA-IIIB NSCLC (IASLC 8th edition).
2. Deemed resectable by MDT.
3. EGFR/ALK wild-type (non-squamous patients; squamous patients exempt).
4. ECOG PS 0-1.
5. Adequate organ function (neutrophils ≥1.5×10⁹/L, platelets ≥100×10⁹/L, Hb >9 g/dL, Cr ≤1.5×ULN, AST/ALT ≤3×ULN).
6. Measurable lesions (RECIST 1.1).

Exclusion Criteria:

1. Active autoimmune diseases (exceptions: vitiligo, type I diabetes, stable hypothyroidism).
2. Systemic corticosteroids (>10 mg prednisone equivalent/day) within 14 days.
3. Grade 3-4 interstitial lung disease.
4. Concurrent malignancies requiring treatment.
5. Prior anti-PD-1/PD-L1/CTLA-4 therapy.
6. Active HBV/HCV, HIV/AIDS, or pregnancy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Estimated)
Dates: Start 2025-05-10 (Actual); Primary Completion 2028-05-10 (Estimated); Study Completion 2030-05-10 (Estimated)

PRIMARY OUTCOMES:
MPR | From date of enrollment until one month after resection
  MPR is defined as ≤10% residual viable tumor in the resected specimen

SECONDARY OUTCOMES:
R0 resection rate | From date of enrollment to an average of 18 weeks after the first dose
  defined as the percentage of patients that undergo R0 surgical resection after neoadjuvant treatment
pCR rate | From date of enrollment until one month after resection
  PCR rate is defined the percentage of patients with no residual viable tumor in the resected specimen
24-month EFS | 36 months following initial treatment
  24-month event-free survival rate in ITT population, defined as the interval between the start of neoadjuvant treatment and any progression of disease precluding surgical resection, progression of disease in the absence of surgery, progression or recurrence after surgery, or death from any cause, whichever occurred first

OTHER OUTCOMES:
Efficacy and safety comparisons between 2-cycle vs. >2-cycle groups | 3 months following resection
  Efficacy (MPR, pCR [percentages]) and safety (TRAEs [percentage]) comparisons between 2-cycle vs. >2-cycle groups.

CONTACTS AND LOCATIONS:
Overall Officials: Ting Zhou, Study Chair — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No